CLINICAL TRIAL: NCT05547542
Title: A Phase 1, Open-label Trial to Evaluate Target Occupancy of CVL-354 at Kappa Opioid and Mu Opioid Receptors in Brain Following Single Oral Doses in Healthy Participants Using Positron Emission Tomography
Brief Title: Positron Emission Tomography (PET) Trial to Evaluate Target Occupancy of CVL-354 at Kappa and Mu Opioid Receptors in Brain Following Oral Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL-354-1002; 4UH3DA052166-02 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder
Keywords: Healthy adult participants
MeSH Terms: conditions — Opioid-Related Disorders | interventions — 3-chloro-4-(4-((2-(3-pyridyl)pyrrolidin-1-yl)methyl)phenoxy)benzamide; carfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Kappa Opioid Receptor (KOR) Cohort (Experimental): Participants will receive single dose of CVL-354, 25 mg, orally, on Day 1 along with [11C]-LY2795050, intravenous (IV) bolus injection of up to 20 millicurie (mCi) before the baseline and post-dose PET scans.
  Based on the KOR receptor occupancy (RO) results from this cohort, dosing may be explored further in subsequent cohorts.
  Interventions: Drug: CVL-354; Drug: [11C]-LY2795050
- Part B: Mu Opioid Receptor (MOR) Cohort (Experimental): Part B will commence after Part A cohort is completed. Participants will receive single dose of CVL-354 150 mg, orally, on Day 1 along with [11C]-carfentanil, IV bolus injection of up to 20 mCi before the baseline and post-dose PET scans.
  Based on the MOR RO results from this cohort, dosing may be explored further in subsequent cohorts.
  Interventions: Drug: CVL-354; Drug: [11C]-carfentanil

INTERVENTIONS:
Drug: CVL-354 — Oral solution/capsule
Drug: [11C]-LY2795050 — IV injection
  Arms: Part A: Kappa Opioid Receptor (KOR) Cohort
Drug: [11C]-carfentanil — IV injection
  Arms: Part B: Mu Opioid Receptor (MOR) Cohort

SUMMARY:
The primary purpose of this study is to assess the target occupancy at kappa and mu opioid receptors in the brain after single oral doses of CVL-354 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Women of nonchildbearing potential and men 18 to 55 years, inclusive, at the time of signing the informed consent form (ICF).
2. Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
3. Body mass index of 18.5 to 32.0 kilograms per square meter (kg/m^2), inclusive, and total body weight >50 kg (110 pounds [lb]) at Screening.
4. Sexually active men with a pregnant or nonpregnant partner of childbearing potential must agree to comply with the following contraception requirements during the trial and for 7 days after the last dose of investigational medicinal product (IMP):

   • Use condom or remain abstinent. In addition, male participants should not donate sperm for a minimum of 7 days following the last dose of IMP.
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
6. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus), malignancy (except for basal cell carcinoma of the skin and cervical carcinoma in situ, at the discretion of the investigator), hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

   * Suicidal Ideation Item 3 (Active Suicidal Ideation with Any Methods [Not Plan] without Intent to Act)
   * Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan)
   * Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent)
   * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, Preparatory Acts or Behavior) "Yes" responses for any of the following items on the C-SSRS (within past 12 months):
   * Suicidal Ideation Item 1 (Wish to be Dead)
   * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts) Serious risk of suicide in the opinion of the investigator is also exclusionary.
3. History of substance or alcohol-use disorder (excluding nicotine or caffeine) as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria within 12 months prior to signing the ICF.
4. Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, uncomplicated appendectomy, and cholecystectomy.
5. Receipt of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccination or booster within 7 days of planned dosing. In addition, participants who plan to receive SARS-CoV-2 vaccination or booster while participating in the trial or for a minimum of 7 days (to cover at least 5 half-lives of IMP) after the last dose of IMP will be excluded.
6. Have recently been diagnosed with symptomatic coronavirus disease-2019 (COVID-19) or test positive (i.e., using polymerase chain reaction (PCR) or rapid antigen test) for COVID-19 within 30 days prior to signing the ICF.
7. Use of prohibited medication prior to randomization or likely to require prohibited concomitant therapy (e.g., prescription and over-the-counter medications, herbal medications, vitamins, and supplements) during the trial.
8. Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
9. Positive drug screen (including cotinine and tetrahydrocannabinol [THC]) or a positive test for alcohol.
10. Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 × upper limit of normal (ULN).
    * Total bilirubin >1.5 × ULN. If Gilbert's syndrome is suspected, total bilirubin >1.5 × ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.
11. Estimated glomerular filtration rate <90 milliliters per minute (mL/min)/1.73 m^2, as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) 2021 equation at the Screening Visit or Check-in (Day -1).

Note: Other protocol-defined Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Kappa Opioid Receptor Occupancy in the Brain Following Single Oral Doses of CVL-354 in Healthy Adult Participants | Day 1
Mu Opioid Receptor Occupancy in the Brain Following Single Oral Doses of CVL-354 in Healthy Adult Participants | Day 1

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to 18 days
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Results | Up to Day 2
Number of Participants With Clinically Significant Changes in Vital Sign Measurements | Up to Day 2
Number of Participants Clinically Significant Changes in Clinical Laboratory Assessments | Up to Day 2
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 2
Number of Participants With Suicidal Ideation and Behavior Assessed Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 2
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.
Maximum Observed Plasma Concentration (Cmax) of CVL-354 During Scan | Day 1 (1.25, 2.0, and 2.75 hours post dose)
Area Under the Plasma Concentration-time Curve (AUC) of CVL-354 for Scan Duration | Day 1 (1.25, 2.0, and 2.75 hours post dose)
Average Plasma Concentration (Cavg) of CVL-354 for Scan Duration | Day 1 (1.25, 2.0, and 2.75 hours post dose)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New Haven, Connecticut, New Haven, Connecticut
  - Yale PET Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No